CLINICAL TRIAL: NCT02823626
Title: High-dose Aldosterone Antagonist for Acute Decompensated Heart Failure
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Relypsa, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HSC20160252H
Record Dates: First submitted 2016-06-27; First posted 2016-07-06 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2018-04

CONDITIONS: Acute Decompensated Heart Failure
MeSH Terms: interventions — Spironolactone; patiromer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intervention: Spironolactone and patiromer
  Interventions: Drug: Spironolactone and patiromer

INTERVENTIONS:
Drug: Spironolactone and patiromer — High dose spironolactone with or without patiromer based on the patient's baseline potassium
  Other Names: Aldactone and veltassa

SUMMARY:
Primary Aims

1. Evaluate the safety of high-dose spironolactone in combination of patiromer in acute decompensated heart failure patients.
2. Evaluate the efficacy of high-dose spironolactone in combination of patiromer in causing volume loss and symptom relief in patients with ADHF treated with high-dose spironolactone.

Secondary Aims

1: Evaluate the effect of high-dose spironolactone on urinary sodium excretion and renal function.

DETAILED DESCRIPTION:
Step-by-Step Methods:

Pre-screening: Patients meeting the inclusion and exclusion criteria will be approached to participate in the study. Informed consent will be taken at this time. These patients will receive intravenous loop diuretic per the discretion of treating physician and will be closely followed for weight loss and symptoms relief.

Screening: The patients who don't respond as measured by symptoms relief or <0.5 kg weight loss/day

1. Despite furosemide ≥ 160 mg IV total daily dose or equivalent dose of torsemide or bumetanide. (1 mg bumetanide = 10 mg torsemide = 20 mg furosemide). OR
2. After 48 hours irrespective of diuretic dose.

will be considered for the study intervention. Patients who have not participated in the pre-screening phase and do not respond adequately to furosemide >160 mg iv daily dose will directly be enrolled into active intervention part of the study.

Intervention (High-Dose Spironolactone + Patiromer): Patients will be initiated on spironolactone 100 mg orally once daily along with patiromer 8.4 gm orally (if serum K >4.3 meq/L). The dose of loop diuretic will stay same during rest of the study period. On day 2, the dose of spironolactone will be titrated to 200 mg orally once a day depending on the diuretic response and lab results. Serum potassium will be monitored twice a day. The dose of patiromer will be increased to 16.8 gm in patients with potassium levels exceeding 5.5 meq/L; or it will be held for serum K <4.3 mEq/L. Treatment will continue till patients achieve euvolemia or get discharged. Euvolemia is defined as resolution of symptoms and signs of volume overload.

Patients will be followed till achievement of euvolemia or discharge. Daily assessment will be done for symptoms, and signs of volume overload including shortness of breath, orthopnea, paroxysmal nocturnal dyspnea, abdominal bloating, lower extremity edema, JVD, and body weight changes. Serum chemistry will be assessed twice a day and urine electrolytes once a day. Neurohormonal analysis will be done at the pre-screening, initiation of active intervention and at the end of the study duration.

Primary Safety Endpoints:

1. Incidence of hyperkalemia as defined by serum K >5.5 meq/day.
2. Renal function: assessed by daily serum creatinine

Primary Efficacy Endpoints:

1. Weight loss: using same calibrated scale every day in hospital gown.
2. Symptom relief: assessed using a 5-point Likert scale describing magnitude of shortness of breath while the patient is in the supine position.

ELIGIBILITY:
Inclusion Criteria:

1. More than18 years old
2. Hospitalized with history of chronic heart failure and at least one symptom (dyspnea, orthopnea or edema) and one sign (rales, peripheral edema, ascites, or radiographic pulmonary edema or pleural effusion)
3. Use of loop diuretics
4. Women of child bearing age with negative urine pregnancy test

Exclusion Criteria:

1. Acute coronary syndrome
2. Patients with a baseline eGFR < 30 ml/min by MDRD equation
3. Baseline potassium concentration ≥ 5.5 mEq/L
4. Requirement for intravenous vasodilators or inotropic agents
5. Systemic infection
6. Patients with concomitant end-stage liver disease
7. Hemodynamically significant uncorrected valvular disease
8. Patients with pulmonary embolism
9. Patients with high output heart failure
10. Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will have been hospitalized with a diagnosis of chronic heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2016-09; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Weight loss | up to 10 days
  Improved swelling and shortness of breath suggestive of volume loss
symptoms relief | up to 10 days
  Improved swelling and shortness of breath suggestive of volume loss

SECONDARY OUTCOMES:
Hypo- or hyperkalemia | up to 10 days
  Serum potassium <3.5 or >5.5 meq/l
Urinary FENa and Urinary Na/K ratio | Up to 10 days
  to measure the sodium loss

CONTACTS AND LOCATIONS:
Overall Officials: Shweta Bansal, Principal Investigator — UT Health San Antonio
Locations (1):
- Shweta Bansal, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT02823626/Prot_SAP_000.pdf